CLINICAL TRIAL: NCT05050851
Title: Nutritional Parameters and Other Risk Factors Affecting Severity of Pneumonia in Children Under Five Years in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Omar Mahmoud Said, Resident at Assiut University children hospital, Assiut University
Other Study IDs: AOMSaid
Record Dates: First submitted 2020-09-21; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Hypoalbuminemia; Stunted Growth; Anemia, Iron Deficiency
Keywords: Pneumonia, nutrition, blood tests, body mass index
MeSH Terms: conditions — Hypoalbuminemia; Growth Disorders; Anemia, Iron-Deficiency; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Measurement of nutritional parameters in children with pneumonia — measurement of Body Mass Index, head circumference, weight, length

SUMMARY:
Decrease mortality rate resulting from pneumonia

DETAILED DESCRIPTION:
Recruiting patients with pneumonia admitted at Assiut University hospital . Then assessment of their condition and severity of pneumonia by examination and X-ray chest . After that, we aim at assessment their nutrition status and it's effect on severity of pneumonia. So we aim to investigate them by CBC, Albumin, CRP and CXR and correlate these parameters with the severity of pneumonia to assess the impact of nutrition on outcome of chest infections

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pneumonia on day 1 of hospital admission.

Exclusion Criteria:

* patients with cardiac diseases
* patients with immune deficiency disorders

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children admitted at Assiut university children hospital below five years with diagnosis of pneumonia on admission.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
ratio of body mass index in patients with pneumonia | Day 1 assessment on hospital admission
  we calculate height of patients in metres and weight in Kg then we divide the weight over the height square to get the body mass index

SECONDARY OUTCOMES:
Concentration of Albumin in patients with pneumonia in g/dl | Day 1 assessment on hospital admission
  blood samlpe will be taken for measuring Albumin level
Hemoglobin level in patients with pnemonia in g/dl | Day 1 assessment on hospital admission
  blood samlpe will be taken for measuring hemoglobin level

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be available to others apart from me as data collector